CLINICAL TRIAL: NCT04920305
Title: Clinical Study on the Effect of Phosphatidylserine on Cognitive Function Improvement in the Elderly
Brief Title: Phosphatidylserine Improves Cognitive Function in the Elderly
Acronym: PICFITE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Air Force Military Medical University, China (Other); Fengdong New Town Elderlywelfare Service Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJTU1AF2021LSY-200
Record Dates: First submitted 2021-05-21; First posted 2021-06-09 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2021-05

CONDITIONS: Aging
Keywords: Aging; Phosphatide; Cognitive
MeSH Terms: interventions — Phosphatidylserines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phosphatidylserine group (Experimental): subjects in the treatment group oral the PS (600mg/d, q.d.) for 6 months.
  Interventions: Dietary Supplement: Phosphatidylserine
- Bean powder group (Placebo Comparator): Subjects in the control group were given a placebo, which was the same shape of bean powder(600mg/d, q.d.) for 6 months.
  Interventions: Dietary Supplement: Bean powder

INTERVENTIONS:
Dietary Supplement: Phosphatidylserine — subjects in the treatment group oral the PS (600mg/d, q.d.) for 6 months.
  Arms: Phosphatidylserine group
Dietary Supplement: Bean powder — Subjects in the control group were given a placebo, which was the same shape of bean powder(600mg/d, q.d.).
  Arms: Bean powder group

SUMMARY:
Cognitive decline is a common symptom of aging, and age-related cognitive impairments are considered normal or inevitable, especially in people over 60, whose memory is more likely to be affected by age. As life expectancy has increased, the number of people with age-related cognitive impairment has also increased. The improvement or slowing of cognitive impairment has received more attention. Phosphatide is a naturally occurring Phosphatide, but it is the main acidic phospholipid in the brain. Phosphatidylserine (PS) is a phospholipid that regulates the function of key proteins in cell membranes and can improve brain function and repair brain damage. PS is thought to enhance neuronal membrane function, which in turn enhances cognitive function. However, there are few studies on the effect of PS on human cognitive function, especially on the elderly, and the results are inconsistent. In this study, people aged 60-70 were given PS intervention for 6 months. Montreal Cognitive Assessment (MOCA) and Mini-Mental State Examination.MMSE) and head MRI are used to evaluate the cognitive function of the subjects before and after the intervention to observe the influence of PS on the cognitive function of the elderly, which is of certain significance for the accurate assessment of the cognitive function of the elderly population and the improvement of the cognitive function of the elderly.

DETAILED DESCRIPTION:
This is a randomized, controlled, double-blind clinical trial, in which 100 subjects were randomly assigned to the treatment group and the control group 1:1 by computer generated random numbers. Before start of the study, all the subjects underwent the first magnetic resonance (MR) and electroencephalogram (EEG) data collection. The working memory capacity of subjects in the N-back paradigm was measured (collected during the N-back task in the EEG test), and the cognition was measured by MOCA and MMSE. After the first data collection was completed, subjects in the treatment group oral the PS (600mg/d, q.d.) for 6 months. Subjects in the control group were given a placebo, which was the same shape of bean powder(600mg/d, q.d.). Under the supervision of nurses, all subjects took the additive at regular times daily. At the end of the 6-month additive trial, all subjects underwent a second MR and EEG data acquisition, as well as measurements of working memory capacity and cognition.

ELIGIBILITY:
Inclusion Criteria:

- Age 60 to 70, gender is not limited.

Exclusion Criteria:

* Delirium, confusion, confusion of consciousness.
* Alzheimer's disease, Parkinson's disease, stroke, cerebral hemorrhage, brain tumor, hydrocephalus.
* Viral, fungal, and syphilis infections.
* Sufferers from cerebrovascular disease (as demonstrated by a Hachinski ischemic score, or neuroimaging test).
* Repeated mild head trauma, or head trauma resulting in loss of consciousness (more than 1h).
* Depression, mania, and other mental disorders.
* Alcoholism and drug dependence.
* The following diseases may lead to mental retardation:

Kidney disease, respiratory system disease, heart disease, liver disease, uncontrolled diabetes, endocrine, metabolic, blood disease, malignant disease, more than 2 years have not been relieved.

* Taken any medication that may cause psychosis or affect intelligence in the past 1 month.
* known allergy to phosphatidylserine or related ingredients.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of functional connectivity, points . | 1 Year
  the strength of functional connectivity, from 0 to 1

SECONDARY OUTCOMES:
The change of point in Montreal Cognitive Assessment (MoCA) test | 1 Year
  MOCA scale from 0 to 30, higher score means higher cognitive ability
The change of point in Mini-mental State Examination (MMSE) test, points. | 1 Year
  MMSE scale from 0 to 30, higher score means higher cognitive ability
The change of working memory test, points. | 1Year.
  The computer program to test memory ability, scale from 0 to 100, higher score means higher memory ability

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Li, Dr., Study Director — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- Fengdong New City Service Center for the Elderly, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No